CLINICAL TRIAL: NCT01612312
Title: Thrombus Aspiration in ThrOmbus Containing culpRiT Lesions in Non-ST-Elevation Myocardial Infarction (TATORT-NSTEMI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Holger Thiele, Co-Director, Department of Internal Medicine/Cardiology, Heart Center Leipzig, University of Leipzig, Germany, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 070-11-07032011
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Non-ST-elevation Myocardial Infarction
Keywords: Non-ST-elevation myocardial infarction; thrombectomy; magnetic resonance imaging; microvascular obstruction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thrombectomy (Active Comparator)
  Interventions: Procedure: Thrombectomy
- Standard percutaneous coronary intervention (Other): In the standard percutaneous coronary intervention (PCI) group, patients will be treated by conventional PCI according to local practice without thrombectomy.
  Interventions: Procedure: Standard percutaneous coronary intervention

INTERVENTIONS:
Procedure: Thrombectomy — Manual thrombectomy will be performed in the thrombus aspiration group using an aspiration catheter utilized in daily clinical routine (Eliminate, Terumo Europe, Leuven, Belgium). In the standard PCI group, patients will be treated by conventional PCI according to local practice without thrombectomy.
  Arms: Thrombectomy
Procedure: Standard percutaneous coronary intervention — In the standard percutaneous coronary intervention (PCI) group, patients will be treated by conventional PCI according to local practice without thrombectomy.
  Arms: Standard percutaneous coronary intervention

SUMMARY:
Whereas thrombus aspiration in patients with ST-elevation myocardial infarction (STEMI) is recommended by current guidelines, there are insufficient data to unequivocally support thrombectomy in patients with non-STEMI (NSTEMI). The Thrombus Aspiration in ThrOmbus containing culpRiT lesions in Non-ST-Elevation Myocardial Infarction (TATORT-NSTEMI) trial is a 400 patient, prospective, controlled, multicenter, randomized, open-label trial. The hypothesis is that under the background of early revascularization, adjunctive thrombectomy in comparison to conventional percutaneous coronary intervention (PCI) alone leads to less microvascular obstruction (MO) assessed by cardiac magnetic resonance imaging (CMR) in patients with NSTEMI. Patients will be randomized in a 1:1 fashion to one of the two treatment arms. The primary endpoint is the extent of MO assessed by CMR. Secondary endpoints include infarct size and myocardial salvage assessed by CMR, enzymatic infarct size as well as angiographic parameters, such as Thrombolysis in Myocardial Infarction-flow post-PCI and myocardial blush grade. Furthermore, clinical endpoints including death, myocardial reinfarction, target vessel revascularization and new congestive heart failure will be recorded at 6 and 12 months. Safety will be assessed by bleeding and stroke. In summary, the TATORT-NSTEMI trial has been designed to test the hypothesis that thrombectomy will improve myocardial perfusion in patients with NSTEMI and relevant thrombus burden in the culprit vessel reperfused by early PCI.

ELIGIBILITY:
Inclusion Criteria:

* ischemic symptoms such as angina pectoris >20 minutes
* occurrence of last symptoms <72 h before randomization
* cardiac troponin T or I levels above the 99th percentile
* culprit lesion containing thrombus (TIMI-thrombus grade 2-5 within the lesion) and intended early PCI

Exclusion Criteria:

* cardiogenic shock
* STEMI
* no identifiable culprit lesion or a TIMI-thrombus grade <2
* coronary morphology ineligible for thrombectomy (e.g. very tortuous vessels, severe calcification)
* indication for acute bypass surgery
* age <18 and >90 years
* contraindications for treatment with heparin, aspirin or thienopyridines
* pregnancy
* current participation in another clinical study
* co-morbidity with limited life expectancy <6 months
* contraindications to CMR at study entry

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Extent of late microvascular obstruction assessed by cardiac magnetic resonance imaging (CMR) | CMR performed within day 1 to 4 after randomization

SECONDARY OUTCOMES:
Infarct size assessed by cardiac magnetic resonance imaging (CMR) | CMR performed within day 1 to 4 after randomization
Myocardial salvage assessed by cardiac magnetic resonance imaging (CMR) | CMR performed within day 1 to 4 after randomization
Left ventricular ejection fraction assessed by cardiac magnetic resonance imaging (CMR) | CMR performed within day 1 to 4 after randomization
Thrombolysis in Myocardial Infarction (TIMI)-flow post-PCI | Immediately after percutaneous coronary intervention
Myocardial blush grade | Immediately after percutaneous coronary intervention
Troponin T | 24 and 48 hours after randomization
Combined clinical endpoint | Follow-up performed at 6, 12 and approximately 60 months after randomization
  Occurence of a combined clinical endpoint including death, re-infarction, target vessel revascularization and congestive heart failure will be recorded. Clinical outcome will be assessed by a telephone interview at 6 and 12 months. Any clinical event will be verified by hospital or general practitioner records.
Assessment of quality of life | 6, 12 and approximately 60 months after randomization
Stroke and bleeding | Participants will be followed for the duration of hospital stay (an expected average of 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Heart Center Leipzig, University of Leipzig, Germany
Locations (7):
- Germany (7):
  - Zentralklinik Bad Berka, Bad Berka
  - Unfallkrankenhaus Berlin, Berlin
  - Klinikum Frankfurt/Oder, Frankfurt (Oder)
  - University of Saarland, Campus Homburg/Saar, Homburg
  - University of Leipzig, Leipzig
  - Institut für Herzinfarktforschung, Ludwigshafen
  - University of Tübingen, Tübingen

REFERENCES:
- [Derived] Lange T, Backhaus SJ, Schulz A, Evertz R, Kowallick JT, Bigalke B, Hasenfuss G, Thiele H, Stiermaier T, Eitel I, Schuster A. Cardiovascular magnetic resonance-derived left atrioventricular coupling index and major adverse cardiac events in patients following acute myocardial infarction. J Cardiovasc Magn Reson. 2023 Apr 13;25(1):24. doi: 10.1186/s12968-023-00929-w. PMID 37046343
- [Derived] Backhaus SJ, Rosel SF, Stiermaier T, Schmidt-Rimpler J, Evertz R, Schulz A, Lange T, Kowallick JT, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Eitel I, Schuster A. Left-atrial long-axis shortening allows effective quantification of atrial function and optimized risk prediction following acute myocardial infarction. Eur Heart J Open. 2022 Aug 12;2(5):oeac053. doi: 10.1093/ehjopen/oeac053. eCollection 2022 Sep. PMID 36268539
- [Derived] Backhaus SJ, Aldehayat H, Kowallick JT, Evertz R, Lange T, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Stiermaier T, Eitel I, Schuster A. Artificial intelligence fully automated myocardial strain quantification for risk stratification following acute myocardial infarction. Sci Rep. 2022 Jul 18;12(1):12220. doi: 10.1038/s41598-022-16228-w. PMID 35851282
- [Derived] Lange T, Stiermaier T, Backhaus SJ, Boom PC, Kowallick JT, de Waha-Thiele S, Lotz J, Kutty S, Bigalke B, Gutberlet M, Feistritzer HJ, Desch S, Hasenfuss G, Thiele H, Eitel I, Schuster A. Functional and prognostic implications of cardiac magnetic resonance feature tracking-derived remote myocardial strain analyses in patients following acute myocardial infarction. Clin Res Cardiol. 2021 Feb;110(2):270-280. doi: 10.1007/s00392-020-01747-1. Epub 2020 Oct 20. PMID 33083869
- [Derived] Schuster A, Lange T, Backhaus SJ, Strohmeyer C, Boom PC, Matz J, Kowallick JT, Lotz J, Steinmetz M, Kutty S, Bigalke B, Gutberlet M, de Waha-Thiele S, Desch S, Hasenfuss G, Thiele H, Stiermaier T, Eitel I. Fully Automated Cardiac Assessment for Diagnostic and Prognostic Stratification Following Myocardial Infarction. J Am Heart Assoc. 2020 Sep 15;9(18):e016612. doi: 10.1161/JAHA.120.016612. Epub 2020 Sep 2. PMID 32873121
- [Derived] Backhaus SJ, Kowallick JT, Stiermaier T, Lange T, Navarra JL, Koschalka A, Evertz R, Lotz J, Kutty S, Hasenfuss G, Gutberlet M, Thiele H, Eitel I, Schuster A. Cardiac Magnetic Resonance Myocardial Feature Tracking for Optimized Risk Assessment After Acute Myocardial Infarction in Patients With Type 2 Diabetes. Diabetes. 2020 Jul;69(7):1540-1548. doi: 10.2337/db20-0001. Epub 2020 Apr 24. PMID 32335515
- [Derived] Feistritzer HJ, Meyer-Saraei R, Lober C, Bohm M, Scheller B, Lauer B, Geisler T, Gawaz M, Bruch L, Klein N, Zeymer U, Eitel I, Jobs A, Freund A, Desch S, de Waha-Thiele S, Thiele H. Long-term outcome after thrombus aspiration in non-ST-elevation myocardial infarction: results from the TATORT-NSTEMI trial : Thrombus aspiration in acute myocardial infarction. Clin Res Cardiol. 2020 Oct;109(10):1223-1231. doi: 10.1007/s00392-020-01613-0. Epub 2020 Feb 6. PMID 32030497
- [Derived] Schuster A, Backhaus SJ, Stiermaier T, Kowallick JT, Stulle A, Koschalka A, Lotz J, Kutty S, Bigalke B, Gutberlet M, Hasenfuss G, Thiele H, Eitel I. Fast manual long-axis strain assessment provides optimized cardiovascular event prediction following myocardial infarction. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1262-1270. doi: 10.1093/ehjci/jez077. PMID 31329854
- [Derived] Backhaus SJ, Kowallick JT, Stiermaier T, Lange T, Koschalka A, Navarra JL, Lotz J, Kutty S, Bigalke B, Gutberlet M, Feistritzer HJ, Hasenfuss G, Thiele H, Schuster A, Eitel I. Culprit vessel-related myocardial mechanics and prognostic implications following acute myocardial infarction. Clin Res Cardiol. 2020 Mar;109(3):339-349. doi: 10.1007/s00392-019-01514-x. Epub 2019 Jul 5. PMID 31278521
- [Derived] Thiele H, de Waha S, Zeymer U, Desch S, Scheller B, Lauer B, Geisler T, Gawaz M, Gunkel O, Bruch L, Klein N, Pfeiffer D, Schuler G, Eitel I. Effect of aspiration thrombectomy on microvascular obstruction in NSTEMI patients: the TATORT-NSTEMI trial. J Am Coll Cardiol. 2014 Sep 16;64(11):1117-24. doi: 10.1016/j.jacc.2014.05.064. PMID 25212646
- [Derived] de Waha S, Eitel I, Desch S, Scheller B, Bohm M, Lauer B, Gawaz M, Geisler T, Gunkel O, Bruch L, Klein N, Pfeiffer D, Schuler G, Zeymer U, Thiele H. Thrombus Aspiration in ThrOmbus containing culpRiT lesions in Non-ST-Elevation Myocardial Infarction (TATORT-NSTEMI): study protocol for a randomized controlled trial. Trials. 2013 Apr 25;14:110. doi: 10.1186/1745-6215-14-110. PMID 23782681